CLINICAL TRIAL: NCT04566289
Title: Observational Registry to Evaluate Real World Usage of PiCSO Impulse System in STEMI Patients as Part of Post-marketing Surveillance
Acronym: PiCSO-AMI-IV
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated due to lack of financing
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: MIR-CIP 0004
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-08

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Anterior MI
Keywords: PiCSO; PiCSO Impulse System
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PiCSO treatment group: PiCSO treatment as per IFU
  Interventions: Device: PiCSO

INTERVENTIONS:
Device: PiCSO — Percutaneous coronary intervention
  Other Names: PCI

SUMMARY:
A prospective, multicenter, single-arm, open label registry of commercially treated patients with PiCSO Impulse System.

DETAILED DESCRIPTION:
This is a observational registry study. Patients with an ST-segment elevated anterior infarct eligible for PCI and commercial PiCSO treatment will be invited to participate in the PiCSO-AMI-IV study. After having given consent as per approved ethics committee requirements, the PCI of the culprit vessel should be performed per standard practices. After blood flow restoration, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS to start the PiCSO therapy. After the procedure the patient will be followed for safety assessments at 30 days, 6 months, 1 year, 2 year and 3 years post index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Culprit lesion in proximal or mid LAD
3. ST-segment elevation
4. Pre-PCI TIMI flow 0 or 1.
5. Symptoms onset time consistent with myocardial ischemia (e.g. persistent chest pain, shortness of breath, nausea/vomiting, fatigue, palpitations or syncope) ≤ 12 h.
6. Patient is deemed eligible for PCI
7. Consent as per approved national ethical committee specific requirements prior to the procedure.

Exclusion Criteria:

1. Patients with contraindications to percutaneous insertion or angiography
2. Patients with implants or foreign bodies in the coronary sinus
3. Known allergy to polyurethanes, PET or stainless steel
4. Known pregnancy or breast feeding
5. Known pericardial effusion or cardiac tamponade
6. Known central hemodynamically relevant left/right shunt
7. Patients with symptom onset > 12 hours
8. Patients with previous CABG
9. Patients with a history of stroke, TIA or reversible ischemic neurological deficit within last 6 month.
10. Patients with coagulopathy
11. Patients under judicial protection, legal guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects presenting with acute myocardial infarction, pre-PCI TIMI flow 0 or 1 and symptom duration ≤ 12 h who are eligible for primary percutaneous coronary intervention as per IFU.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Device Effect (ADE) rate at 30 days post index procedure PCI | 30 days
  Adverse Device Effect (ADE) rate at 30 days post index procedure PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Dresden GmbH Universitätsklinik an der TU Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided